

# Clinical Development

# ETB115/eltrombopag/Promacta®/Revolade®

### CETB115E2403 / NCT02998645

SOAR, Interventional phase II single-arm study to assess efficacy and safety of eltrombopag combined with cyclosporine as first line therapy in adult patients with severe acquired aplastic anemia

Statistical Analysis Plan (SAP) - Amendment 4

Author: (Trial statistician)

Document type: SAP Documentation

Document status: Final v1.0

Release date: 23- Jun-2022

Number of pages: 44

Property of Novartis
For business use only
May not be used, divulged, published or otherwise disclosed
without the consent of Novartis

# Document History – Changes compared to previous final version of SAP

| Date | Time<br>point | Reason for update | Outcome for update | Section and title impacted (Current) |
|---|---|---|---|---|
| 28-Mar-2017 | Prior<br>FPFV | N/A – Initial<br>version | N/A | N/A |
| 26-Oct-2017<br>Amendment | After<br>FPFV | Incorporate changes from protocol | Further clarification on endpoints and sample size calculation. | Sec 1, 2 and 4 |
| 1 | | amendment 1 dated<br>17-May-2017 | Only overall survival tables will<br>be summarised by responder<br>status | |
| 26-Jul-2019<br>Amendment | After 31 | Incorporate changes | Updated endpoints | Sec 1, 2 and 4 |
| 2 | patients<br>enrolled | from protocol<br>amendment 2 dated<br>26-Feb-2019 | Duration of trial shortened from 60 to 24 months | |
| | | | Removal of overall survival and paediatric analyses | |
| 03-Dec-2020<br>Amendment<br>3 | Enrollment complete | Updates after dry run | Clarification on derivation of planned dose intensity. Exclusion of patients from per protocol set based on COVID19 protocol deviations were added. For response derivations if due to COVID19 patient has local instead of central lab result for scheduled visit, these local results will be used. Replaced Race subgroup with Ethnicity subgroup. Updated derivations for clonal evolution. All deaths listing will included patients who died in screening. Updates to PK and biomarker sections. Added sample size characteristics based on 54 enrolled patients. | Sec 1, 2 and 4 |
| 23-Jun-2022<br>Amendment<br>4 | Prior final<br>data base<br>lock | Based on<br>recommendation of<br>steering committee<br>members and<br>comments from the<br>dry run | Information about interim database lock for primary analysis is added. Age categories is changed to <60, >=60. Additional subgroups analysis by age, ethnicity and/or responder status were added for demographic characteristics, overall hematological response, | Sec 1,<br>2.2.6, 2.3.2,<br>2.5.1, 2.5.2, 2.6.1,<br>2.6.2,<br>2.6.5, 2.7.1, 2.9<br>and 4 |

| Date | Time<br>point | Reason for<br>update | Outcome for update | Section and title impacted (Current) |
|---|---|---|---|---|
| | | | transfusion information and relevant AEs. | |
| | | | Sample timing for primary endpoint was clarified. | |
| | | | Clarification on derivation of duration of hematologic response. | |
| | | | Clarification on definition of the start and end dates for the transfusion independence. | |
| | | | Updated PROs text with including information on boxplots. | |

# **Table of contents**

| | Table | of conte | nts | 4 |
|---|---|---|---|---|
| | List o | f abbrevi | ations | 6 |
| 1 | Introd | duction | | 8 |
| | 1.1 | Study d | lesign | 8 |
| | 1.2 | Study o | objectives and endpoints | 9 |
| 2 | Statis | | hods | |
| | 2.1 | Data an | nalysis general information | 11 |
| | | 2.1.1 | Data included in the analysis | 11 |
| | | 2.1.2 | General analysis conventions | 12 |
| | | 2.1.3 | General definitions | 12 |
| | 2.2 | Analys | is sets | 17 |
| | | 2.2.1 | Full Analysis Set | 17 |
| | | 2.2.2 | Safety Set | 17 |
| | | 2.2.3 | Per-Protocol Set | 17 |
| | | 2.2.4 | Pharmacokinetic Analysis Set | 18 |
| | | 2.2.5 | Screening failures | 18 |
| | | 2.2.6 | Subgroups of interest | 18 |
| | 2.3 | Patient | disposition, demographics and other baseline characteristics | 19 |
| | | 2.3.1 | Patient disposition | 19 |
| | | 2.3.2 | Patient demographics and other baseline characteristics | 19 |
| | 2.4 | Treatm | ents (study treatment, concomitant therapies and compliance) | |
| | | 2.4.1 | Study treatment | 20 |
| | | 2.4.2 | Prior, concomitant and post therapies | 20 |
| | | 2.4.3 | Protocol deviations | 20 |
| | | 2.4.4 | Handling of missing values | 21 |
| | 2.5 | Analys | is of the primary objective | 21 |
| | | 2.5.1 | Primary endpoint | 21 |
| | | Handlii | ng of missing values/discontinuations | 22 |
| | | 2.5.2 | Supportive analyses | 22 |
| | 2.6 | Analys | is of secondary efficacy objective(s) | 22 |
| | | 2.6.1 | ORR by 3 months, at 12 months and at 24 months | 22 |
| | | 2.6.2 | Duration of hematologic response | 23 |
| | | 2.6.3 | Relapse rate | 23 |
| | | 2.6.4 | Clonal evolution | 23 |
| | | 265 | Blood (RBC) and platelet transfusions | 24 |

| | 2.7 | Safety a | analyses | 24 |
|---|---|---|---|---|
| | | 2.7.1 | Adverse events (AEs) | 24 |
| | | 2.7.2 | Deaths | 26 |
| | | 2.7.3 | Laboratory data | 26 |
| | | 2.7.4 | Other safety data | 27 |
| | 2.8 | Pharma | cokinetic endpoints | 29 |
| | 2.9 | Patient- | reported outcomes (PROs) | 30 |
| | | 2.9.1 | FACIT-Fatigue and FACT-TH18 (includes FACT-G) | 30 |
| | | | | 31 |
| | | | | 32 |
| | | | | 32 |
| | | | | 32 |
| | | | | 33 |
| | | | | 33 |
| | | | | 34 |
| | 2.11 | Interim | analysis | 35 |
| 3 | Samp | le size ca | lculation | 35 |
| | | 3.1.1 | Bayesian calculus for a binary endpoint | 36 |
| 4 | Chang | ges to pro | otocol specified analyses | 36 |
| 5 | Refere | ences | | 37 |
| 6 | Appei | ndix 1 | | 38 |
| | 6.1 | Imputat | tion rules | 38 |
| | | 6.1.1 | AE, concomitant medication (CM) and safety assessment date | |
| | | | imputation | 38 |
| | | 6.1.2 | Prior therapies date imputation | 39 |
| | 6.2 | Laborat | tory parameters derivations | 39 |
| | 6.3 | Statistic | cal models | 39 |
| | | 6.3.1 | Primary analysis | 39 |
| | | 6.3.2 | Key secondary analysis | 40 |
| | 6.4 | FACIT- | -Fatigue scoring guideline | 40 |
| | 6.5 | FACT- | Th18 and FACT-G scoring guideline | 41 |

### List of abbreviations

AE adverse event

AESI adverse events of special interest

ALP alkaline phosphatase
ALT alanine aminotransferase
ANC absolute neutrophil count
AST aspartate aminotransferase

ATC anatomical therapeutic classification

ATG anti-thymocyte globulin AUC area under the curve

BM bone marrow

CM concomitant medication
CR complete response
CRS case retrieval sheet
CSR clinical study report

CTCAE common terminology criteria for adverse events

CV coefficient of variation
DHP data handling plan
DI dose intensity

DNA deoxyribonucleic acid EC/ECG electrocardiogram

ECOG eastern cooperative oncology group

eCRF electronic case report form

EOT end of treatment

FACIT functional assessment of chronic illness therapy

FAS full analysis set FPFV first patient first visit

GPS global programming & statistical environment

HLGT high level group term
HLT high level term
HR heart rate

IST immunosuppressive therapy

LB laboratory

LLOQ lower limit of quantification LPLV last patient last visit

MedDRA medical dictionary for drug regulatory affairs

NCDS Novartis clinical data standards
NGS next generation sequencing
NMQ Novartis MedDRA queries
ORR overall response rate
PA protocol amendment

PAS pharmacokinetic analysis set PDI planned dose intensity

PDS programming data specifications

PK pharmacokinetics

PNH paroxysmal nocturnal hemoglobinuria

PPS per-protocol set

PR partial response

PRO patient-reported outcomes

PT preferred term

QTcF QT correction Fridericia

RBC red blood cells

RDI relative dose intensity

RT-PCR reverse transcription polymerase chain reaction

SAA severe aplastic anemia
SAE serious adverse event
SAP statistical analysis plan
sd standard deviation

SI international system of units
SMQs standardized MedDRA queries

SOC system organ class TBL total bilirubin

TFLs tables, figures, listings
TPO-R thrombopoietin receptor
ULOQ upper limit of quantification

VS vital signs

### 1 Introduction

This statistical analysis plan (SAP), describes the analyses for the CETB115E2403 study and is based on protocol v02, dated 26-Feb-2019. Enrollment was completed on 11-May-2020 with fifty four (54) adult patients. The interim database lock for the primary analysis was on 09-Dec-2020.

There are 2 planned reporting events:

- 1. The **primary analysis**, was done after all enrolled patients completed **6 months** or discontinued prior to 6 months. A primary clinical study report (CSR) was written.
- 2. The **final analysis** will be done after all patients have completed the study or discontinued early, for the patients responding at 6 months this will be once they have completed **24 months** in the study or discontinued the study prior to 24 months. A final CSR will be written.

The shells for the in-text tables and figures as well as the post-text tables, figures and listings (TFLs) are in the TFL shells document. Programming specifications for datasets, including derivation of variables, are given in the programming data specifications (PDS) document.

All data will be analysed by Novartis using Novartis clinical data standards (NCDS). Analysis data sets and statistical outputs will be produced using the SAS system Version 9.4 or higher (UNIX environment) in the global programming & statistical (GPS) environment

# 1.1 Study design

The study design is shown in Figure 1-1 and Figure 1-2.

This is an interventional, phase II, single-arm, multicenter, open-label, study to investigate the efficacy and safety of the combination of eltrombopag and cyclosporine in treatment-naive adult patients with severe aplastic anemia (SAA) as first line therapy administered for 6 months, with an additional 18 months follow-up for responders for cyclosporine tapering and duration of response until relapse or 24 months whichever is earlier.

At 6 months, **responders** will discontinue eltrombopag and start to taper cyclosporine until 24 months. Responders who are no longer responding at 6 months and **non-responders** will discontinue the treatment and study at 6 months and will be followed-up for 30 days. Responders who relapse prior to 24 months will discontinue cyclosporine and study, and will be followed-up for 30 days.

Responders who relapse and non-responders already in the follow-up under the previous protocol version will be discontinued from the study within 30 days of the approval of the protocol amendment.

The lack of availability of anti-thymocyte globulin (ATG) in several countries has left a large proportion of patients with SAA with limited treatment options and poor outcome. In this context, the combination of cyclosporine and eltrombopag, 2 therapies with different modes of action, is an attractive therapeutic option to address this unmet medical need. Cyclosporine acts as an immunosuppressant and eltrombopag acts as a stimulator of bone marrow progenitor cells.

Fifty (50) patients are planned to be enrolled.

### Figure 1-1 Study design under protocol amendment 1

Under protocol amendment (PA) 1 (4 phases: Treatment 1; Treatment 2; Follow-up; post-treatment follow-up)



Figure 1-2 Study design under protocol amendment 2

Under PA2 (2 phases: Treatment 1 and Treatment 2)



<sup>\*</sup> Follow-up for duration of response until relapse or Month 24 whichever is earlier for responders only who did not relapse prior to Month 6

# 1.2 Study objectives and endpoints

Table 1-1 displays the study objectives and endpoints.

Table 1-1 Objectives and related endpoints

| Objective | Endpoint |
|---|---|
| Primary | |
| To evaluate the efficacy of eltrombopag + cyclosporine as first-line therapy on overall hematologic response (partial and complete response) by 6 months | Overall hematologic response (CR + PR)* rate by 6 months (definition of CR and PR is given as footnote below) |

| 1. Evaluate the effect of eltrombopag + cyclosporine on overall hematologic response (partial and complete response): ■ by 3 months ■ at 12 months ■ at 12 months ■ at 24 months 1. Evaluate the duration of hematologic response (partial and complete response): ■ at 12 months ■ at 24 months 1. To evaluate the duration of hematologic response appropriate and will be reported in a cumulative basis until the cutoff date (LPLV for final analysis) 2. To evaluate the proportion of patients who relapse 4. To evaluate the proportion of patients who relapse 4. To evaluate the clonal evolution to myelodysplasia, paroxysmal nocturnal hemoglobinuria (PNH), and leukemia 5. To evaluate red blood cells (RBC) transfusion independence 6. To evaluate platelet transfusion independence 7. To evaluate the longest interval without a platelet and RBC transfusion 1. To evaluate the effect of Eltrombopag and cyclosporine on patient symptoms and health related quality of life 9. To evaluate the safety and tolerability of eltrombopag + cyclosporine 10. To characterize the PK of eltrombopag when combined to cyclosporine Overall hematologic response (CR + PR)' rate: • by 3 months • at 2 months • at 2 months • at 24 months (responders only) as appropriate and will be responders only a months and 24 months or RBC transfusion in the study Percentage of patients who are RBC transfusion independence defined as no RBC transfusion or at least 56 days Duration of longest interval without a platelet transfusion or at least 28 days Duration of longest interval without a platelet transfusion by 6 months and 24 months. Independence defined as no platelet transfusion by 6 months and 24 months. Or applied to transfusion by 6 months and 24 months. Or applied to transfusion by 6 months and 24 months. Or applied to transfusion by 6 months and 24 months. Or applied to transfusion by 6 months and 24 months. Or applied to transfusion by 6 months and 24 months. Or applied transfusion by 6 months and 24 months. Or applied to transfusion by 6 | Objective | Endpoint |
|---|---|---|
| eyclosporine on overall hematologic response (partial and complete response): • by 3 months • at 12 months • at 24 months The following secondary objectives will be assessed by 6 months and 24 months (responders only) as appropriate and will be reported in a cumulative basis until the cutoff date (LPLV for final analysis) cresponse 2. To evaluate the duration of hematologic response 3. To evaluate the proportion of patients who relapse 4. To evaluate the proportion of patients who relapse 4. To evaluate the clonal evolution to myelodysplasia, paroxysmal nocturnal hemoglobinuria (PNH), and leukemia 5. To evaluate red blood cells (RBC) transfusion independence 6. To evaluate platelet transfusion independence 6. To evaluate the longest interval without a platelet and RBC transfusion independence defined as no RBC transfusion of at least 328 days 7. To evaluate the effect of Eltrombopag and cyclosporine on patient symptoms and health related quality of life 9. To evaluate the safety and tolerability of eltrombopag + cyclosporine 10. To characterize the PK of eltrombopag when combined to evolosporine * by 3 months • at 24 months • at 24 months • at 24 months (responders only) as appropriate at 24 months (responders only) as appropriate and will the cutoff date (LPLV for final analysis) • Time from the date of the first response to the date of first relapse (defined as no longer meeting definition of PR (and not CR) Percentage of patients who relapse Percentage of patients with evolution to myelodysplasia, PNH, and acute leukemia occurring at any time during the study Percentage of patients who are RBC transfusion independence defined as no RBC transfusion for at least 328 days Percentage of patients who are RBC transfusion for at least 328 days Percentage of patients who are platelet transfusion independence defined as no platelet transfusion by 6 months and 24 months Duration of longest interval without a platelet transfusion by 6 months and 24 months Charge in scores from baseline to 6 months | Secondary | Secondary |
| appropriate and will be reported in a cumulative basis until the cutoff date (LPLV for final analysis) 2. To evaluate the duration of hematologic response Time from the date of the first response to the date of first relapse (defined as no longer meeting definition of PR (and not CR) 3. To evaluate the proportion of patients who relapse 4. To evaluate the clonal evolution to myelodysplasia, paroxysmal nocturnal hemoglobinuria (PNH), and leukemia 5. To evaluate red blood cells (RBC) transfusion independence 5. To evaluate platelet transfusion independence 6. To evaluate platelet transfusion independence 7. To evaluate the longest interval without a platelet and RBC transfusion 1. To evaluate the effect of Eltrombopag and cyclosporine on patient symptoms and health related quality of life 9. To evaluate the safety and tolerability of eltrombopag + cyclosporine 10. To characterize the PK of eltrombopag when combined to cyclosporine Time from the date of the first response to the date of first relapse (defined as no longer meeting definition of PR (and not CR) Time from the date of the first response to the date of first relapse (defined as no longer meeting definition of PR (and not CR) Percentage of patients who relapse Percentage of patients who are RBC transfusion independent at least once by 6 months and by 24 months. Independence defined as no RBC transfusion of at least 28 days Duration of longest interval without a platelet transfusion by 6 months and 24 months Change in scores from baseline to 6 months and 24 months on the FACT-G, FACT-TH18, and FACIT-Fatigue scales Safety will be assessed by: • Frequency and severity of AEs, serious AEs (SAEs) based on the Common Terminology Criteria of Adverse Events (CTCAE version 4. 03), and AEs leading to discontinuation, and evaluating changes in laboratory values within 6 months and within 24 months (responders only) • Incidence of adverse events of special interest Plasma PK parameters of eltrombopag at 2 weeks and trough concentrations at 1 mo | cyclosporine on overall hematologic response (partial and complete response): • by 3 months • at 12 months | <ul><li>by 3 months</li><li>at 12 months</li></ul> |
| relapse (defined as no longer meeting definition of PR (and not CR) 3. To evaluate the proportion of patients who relapse 4. To evaluate the clonal evolution to myelodysplasia, paroxysmal nocturnal hemoglobinuria (PNH), and leukemia 5. To evaluate red blood cells (RBC) transfusion independence 6. To evaluate platelet transfusion independence 7. To evaluate platelet transfusion independence 8. To evaluate the longest interval without a platelet and RBC transfusion 9. To evaluate the effect of Eltrombopag and cyclosporine on patient symptoms and health related quality of life 9. To evaluate the safety and tolerability of eltrombopag + cyclosporine 10. To characterize the PK of eltrombopag when combined to cyclosporine relapse (defined as no longer meeting definition of CR) Percentage of patients who relapse Percentage of patients with evolution to myelodysplasia, PNH, and acute leukemia occurring at any time during the study Percentage of patients with evolution to myelodysplasia, PNH, and acute leukemia occurring at any time during the study Percentage of patients with evolution to myelodysplasia, PNH, and acute leukemia occurring at any time during the study Percentage of patients with evolution to myelodysplasia, PNH, and acute leukemia occurring at any time during the study Percentage of patients with evolution to myelodysplasia, PNH, and acute leukemia occurring at any time during the study Percentage of patients with evolution to myelodysplasia, PNH, and acute leukemia occurring at any time during the study Percentage of patients with evolution to myelodysplasia, PNH, and acute leukemia occurring at any time during the study Percentage of patients with evolution to myelodysplasia, PNH, and acute leukemia occurring at any time during the study Percentage of patients with evolution to myelodysplasia, PNH, and acute leukemia occurring at any time during the study Percentage of patients with evolution to myelodysplasia, PNH, and acute leukemia occurring at any time during the study Percent | | |
| relapse 4. To evaluate the clonal evolution to myelodysplasia, paroxysmal nocturnal hemoglobinuria (PNH), and leukemia 5. To evaluate red blood cells (RBC) transfusion independence 6. To evaluate platelet transfusion independence 7. To evaluate the longest interval without a platelet and RBC transfusion 8. To evaluate the effect of Eltrombopag and cyclosporine on patient symptoms and health related quality of life 9. To evaluate the safety and tolerability of eltrombopag + cyclosporine 10. To characterize the PK of eltrombopag when combined to cyclosporine 4. To evaluate the clonal evolution to myelodysplasia, PNH, and acute leukemia occurring at any time during the study Percentage of patients who are RBC transfusion independent at least once by 6 months and by 24 months. Independence defined as no platelet transfusion independence defined as no platelet transfusion of longest interval without a platelet transfusion by 6 months and 24 months Duration of longest interval without a platelet transfusion by 6 months and by 24 months Change in scores from baseline to 6 months and 24 months on the FACT-G, FACT-TH18, and FACIT-Fatigue scales Safety will be assessed by: • Frequency and severity of AEs, serious AEs (SAEs) based on the Common Terminology Criteria of Adverse Events (CTCAE version 4. 03), and AEs leading to discontinuation, and evaluating changes in laboratory values within 6 months and within 24 months (responders only) • Incidence of adverse events of special interest Plasma PK parameters of eltrombopag at 2 weeks and trough concentrations at 1 month, 2 months, 3 month, and | | relapse (defined as no longer meeting definition of PR (and |
| myelodysplasia, paroxysmal nocturnal hemoglobinuria (PNH), and leukemia 5. To evaluate red blood cells (RBC) transfusion independence 6. To evaluate platelet transfusion independence 6. To evaluate platelet transfusion independence 7. To evaluate the longest interval without a platelet and RBC transfusion 8. To evaluate the effect of Eltrombopag and cyclosporine on patient symptoms and health related quality of life 9. To evaluate the safety and tolerability of eltrombopag + cyclosporine 10. To characterize the PK of eltrombopag when combined to cyclosporine PNH, and acute leukemia occurring at any time during the study PRH, and acute leukemia occurring at any time during the study PRH, and acute leukemia occurring at any time during the study Precentage of patients who are RBC transfusion for at least 56 days Percentage of patients who are platelet transfusion independent at least once by 6 months and by 24 months. Independence defined as no platelet transfusion independent at least once by 6 months and by 24 months. Independence defined as no platelet transfusion independent at least once by 6 months and by 24 months. Independence defined as no platelet transfusion independent at least once by 6 months and by 24 months. Independence defined as no platelet transfusion independent at least once by 6 months and by 24 months. Independence defined as no platelet transfusion independence defined as no platelet transfusion independence defined as no platelet transfusion independence defined as no platelet transfusion independence defined as no platelet transfusion of longest interval without a platelet transfusion by 6 months and by 24 months. Change in scores from baseline to 6 months and 24 months on the FACT-G, FACT-TH18, and FACIT-Fatigue scales Safety will be assessed by: • Frequency and severity of AEs, serious AEs (SAEs) based on the Common Terminology Criteria of Adverse Events (CTCAE version 4. 03), and AEs leading to discontinuation, and evaluating changes in laboratory values within 6 month | · | Percentage of patients who relapse |
| independent at least once by 6 months and by 24 months. Independence defined as no RBC transfusion for at least 56 days 6. To evaluate platelet transfusion independence 7. To evaluate the longest interval without a platelet and RBC transfusion 8. To evaluate the effect of Eltrombopag and cyclosporine on patient symptoms and health related quality of life 9. To evaluate the safety and tolerability of eltrombopag + cyclosporine 10. To characterize the PK of eltrombopag when combined to cyclosporine independent at least once by 6 months and by 24 months. Independence defined as no platelet transfusion independent at least once by 6 months and by 24 months. Independence defined as no platelet transfusion for at least 28 days Duration of longest interval without a platelet transfusion by 6 months and 24 months of longest interval without a platelet transfusion by 6 months and 24 months Change in scores from baseline to 6 months and 24 months on the FACT-G, FACT-TH18, and FACIT-Fatigue scales Safety will be assessed by: Frequency and severity of AEs, serious AEs (SAEs) based on the Common Terminology Criteria of Adverse Events (CTCAE version 4. 03), and AEs leading to discontinuation, and evaluating changes in laboratory values within 6 months and within 24 months (responders only) Incidence of adverse events of special interest Plasma PK parameters of eltrombopag at 2 weeks and trough concentrations at 1 month, 2 months, 3 month, and | myelodysplasia, paroxysmal nocturnal | PNH, and acute leukemia occurring at any time during the |
| independence independent at least once by 6 months and by 24 months. Independence defined as no platelet transfusion for at least 28 days 7. To evaluate the longest interval without a platelet and RBC transfusion 8. To evaluate the effect of Eltrombopag and cyclosporine on patient symptoms and health related quality of life 9. To evaluate the safety and tolerability of eltrombopag + cyclosporine 9. To evaluate the safety and tolerability of eltrombopag + cyclosporine 10. To characterize the PK of eltrombopag when combined to cyclosporine independent at least once by 6 months and by 24 months. Independent at least once by 6 months and by 24 months Independent at least once by 6 months and by 24 months Independent at least once by 6 months and by 24 months Independent at least once by 6 months and by 24 months Independent at least once by 6 months and by 24 months Independent at least once by 6 months and better transfusion by 6 months and 24 months Change in scores from baseline to 6 months and 24 months of months and 24 months Change in scores from baseline to 6 months and 24 months of months and 24 months Change in scores from baseline to 6 months and 24 months Change in scores from baseline to 6 months and 24 months Change in scores from baseline to 6 months and 24 | | independent at least once by 6 months and by 24 months. Independence defined as no RBC transfusion for at least |
| by 6 months and 24 months Duration of longest interval with a RBC transfusion by 6 months and by 24 months 8. To evaluate the effect of Eltrombopag and cyclosporine on patient symptoms and health related quality of life 9. To evaluate the safety and tolerability of eltrombopag + cyclosporine Safety will be assessed by: • Frequency and severity of AEs, serious AEs (SAEs) based on the Common Terminology Criteria of Adverse Events (CTCAE version 4. 03), and AEs leading to discontinuation, and evaluating changes in laboratory values within 6 months and within 24 months (responders only) • Incidence of adverse events of special interest Plasma PK parameters of eltrombopag at 2 weeks and trough concentrations at 1 month, 2 months, 3 month, and | | independent at least once by 6 months and by 24 months. Independence defined as no platelet transfusion for at |
| cyclosporine on patient symptoms and health related quality of life 9. To evaluate the safety and tolerability of eltrombopag + cyclosporine Safety will be assessed by: • Frequency and severity of AEs, serious AEs (SAEs) based on the Common Terminology Criteria of Adverse Events (CTCAE version 4. 03), and AEs leading to discontinuation, and evaluating changes in laboratory values within 6 months and within 24 months (responders only) • Incidence of adverse events of special interest Plasma PK parameters of eltrombopag at 2 weeks and trough concentrations at 1 month, 2 months, 3 month, and | • | by 6 months and 24 months Duration of longest interval with a RBC transfusion by |
| <ul> <li>Frequency and severity of AEs, serious AEs (SAEs) based on the Common Terminology Criteria of Adverse Events (CTCAE version 4. 03), and AEs leading to discontinuation, and evaluating changes in laboratory values within 6 months and within 24 months (responders only)</li> <li>Incidence of adverse events of special interest</li> <li>To characterize the PK of eltrombopag when combined to cyclosporine</li> </ul> | cyclosporine on patient symptoms and health | months on the FACT-G, FACT-TH18, and FACIT-Fatigue |
| when combined to cyclosporine trough concentrations at 1 month, 2 months, 3 month, and | , | • Frequency and severity of AEs, serious AEs (SAEs) based on the Common Terminology Criteria of Adverse Events (CTCAE version 4. 03), and AEs leading to discontinuation, and evaluating changes in laboratory values within 6 months and within 24 months (responders only) |
| | | trough concentrations at 1 month, 2 months, 3 month, and |



\*Overall hematologic response = patients with complete response (CR) + patients with partial response (PR) a. Partial response is defined as any two of the following parameters at two consecutive, scheduled visit measurements at least 7 days apart during the study (and not sufficient for CR) and no platelet transfusions within 7 days of platelet measurement (can still be a responder if ANC and reticulocyte measurements are valid):

- Absolute neutrophil count (ANC) ≥ 500/µL
- Platelet count ≥ 20 000/µL
- Reticulocyte count ≥ 60 000/µL (automated)
- b. Complete response is defined as all three parameters meet the following criteria at two consecutive, scheduled visit measurements at least 7 days apart during the study and no platelet transfusions within 7 days of platelet measurement and no RBC transfusion with 14 days of the hemoglobin measurements:
  - Absolute neutrophil count (ANC) ≥ 1 000/µL
  - Platelet count ≥ 100 000/µL
  - Hemoglobin ≥ 10g/dL

Example: At the end of 6 months out of 50 patients enrolled, if 13 patients satisfy the criteria for CR and 3 patients satisfy the criteria for PR, the overall hematologic response will be 13+3=16 patients.

### 2 Statistical methods

### 2.1 Data analysis general information

### 2.1.1 Data included in the analysis

Statistical analyses will be performed using all data collected in the database up to the respective data cut-off dates (last patient last visit (LPLV) for the final analysis). All data with an assessment date or event start date (e.g. vital sign assessment date or start date of an adverse event (AE)) prior to or on the cut-off date will be included in the analysis. Any data collected beyond the cut-off date will not be included in the analysis and will not be used for any derivations.

All events with start date before or on the cut-off date and end date after the cut-off date or missing will be reported as 'ongoing'. For these events, the end date will show as missing in the listings however the earliest of; death date, last contact date or cutoff date will be used in derivations of endpoints as appropriate.

### Withdrawal of Informed Consent

Any data collected in the clinical database after a patient withdraws informed consent from all further participation in the trial, will not be included in the analysis. The date on which a patient withdraws full study consent is recorded in the electronic case report form (eCRF).

### 2.1.2 General analysis conventions

Data from all study centers will be pooled for analyses.

Qualitative data (e.g., gender, race, etc.) will be summarised by absolute and relative frequencies. A missing category will be included where applicable. Percentages will be calculated using the number of patients in the relevant analysis set or subgroup as the denominator.

**Quantitative data** (e.g., age, body weight, etc.) will be summarised by appropriate descriptive statistics (i.e. mean, standard deviation (sd), minimum, 25<sup>th</sup> percentile, median, 75<sup>th</sup> percentile and maximum).

### 2.1.3 General definitions

### Study drug and study treatment

Study drugs refer to the individual drugs used in the study, eltrombopag or cyclosporine.

Study treatment refers to either eltrombopag or cyclosporine or eltrombopag+cyclosporine.

### Date of first administration of study drug

The date of first administration of study drug is derived as the first date when a nonzero dose of study drug is administered. The date of first administration of study drug is also referred to as **start date of study drug**. Start date of study drug is defined for each study drug. For cyclosporine it is irrespective of capsule or solution form.

### Date of last administration of study drug

The date of last administration of study drug is defined as the last date when a nonzero dose of study drug is administered. This date is also referred to as *last date of study drug*. Last date of study drug is defined for each study drug. For cyclosporine it is irrespective of capsule or solution form.

### Date of first administration of study treatment

The date of first administration of study treatment is derived as the first date when a nonzero dose of any component of study treatment is administered.

For example, if the 1<sup>st</sup> dose of eltrombopag is taken on 08-Feb-2017, and 1<sup>st</sup> dose of cyclosporine, is taken on 07-Feb-2017, then the date of first administration of study treatment is 07-Feb-2017. The date of first administration of study treatment is also referred to as *start date of study treatment*.

### Date of last administration of study treatment

The date of last administration of study treatment is derived as the last date when a nonzero dose of any component of study treatment is administered.

For example if the last dose of eltrombopag is taken on 08-Aug-2017, and the last dose of cyclosporine is taken on 07-Aug-2017, then the date of last administration of study treatment is on 08-Aug-2017. This date is also referred to as *last date of study treatment*.

### **Duration of exposure**

The duration of exposure for the **study drugs** will be calculated as:

• Duration of study drug exposure (months) = (last date of study drug) – (first date of study drug) + 1.

The duration of exposure for the **study treatment** will be calculated as:

• Duration of study treatment exposure (months) = (last date of study treatment) – (first date of study treatment) + 1.

If the start or end date of a study drug is missing, the duration will be missing. The durations will include periods of temporary interruption (planned or actual) for any reason.

### **Dose interruption**

An interruption is defined as an actual zero dose on one or more days between two non-zero dosing records.

Note: The last zero dose of a study drug (followed by permanent discontinuation) is not considered as a dose interruption. For the purpose of summarizing interruptions and reasons, in case multiple entries for interruption are entered on consecutive days with different reasons these will be counted as separate interruptions. However, if the reason is the same in these multiple entries on consecutive days, then it will be counted as one interruption.

### **Dose reduction**

A dose reduction is where the prescribed dose is lower than the previous prescribed dose or where the actual dose administered/total daily dose is lower than the prescribed dose. Any dose change to correct a dosing error will not be considered a dose reduction, e.g. if due to a dosing error, a patient receives higher than protocol planned starting dose and moves down to the planned starting dose then this is not counted as a reduction, however if they move directly from a higher than planned starting dose down to a lower than protocol planned starting dose, then this is counted as a reduction.

Note: It is assumed that if there is a dose reduction, then the 'Dose changed' box was ticked on the dose administration eCRF page.

#### Cumulative dose

Cumulative dose of a study treatment is defined as the total dose given during the study treatment exposure and will be summarised for each of the study treatment components (eltrombopag and cyclosporine), respectively.

The **planned cumulative dose** for a study treatment component refers to the total planned dose as per the protocol up to the last date of study drug administration. The planned cumulative dose is not summarised/listed. It is used for relative dose intensity calculations. The **actual cumulative dose** refers to the total actual dose administered, over the duration for which the patient is on the study treatment as documented in the dose administration eCRF.

For continuous dosing, the actual cumulative dose is the sum of the non-zero doses recorded over the dosing period and the planned cumulative dose is the planned starting dose summed over the same dosing period.

For cyclosporine the cumulative dose will be calculated separately for capsules (mg) and solution (mg/ml).

For patients who did not take any drug, the actual cumulative dose is by definition equal to zero for that drug.

### Dose intensity and relative dose intensity

**Dose intensity (DI)** for patients with non-zero duration of exposure is defined as follows:

DI (*dosing unit / unit of time*) = Actual cumulative dose (*dosing unit*) / Duration of exposure (*unit of time*).

```
e.g. DI (mg/day) = (100 \text{ mg/day} * 1050 \text{ days}) / 1080 \text{ days} = 97.2 \text{ mg/day}
```

For patients who did not take any drug the DI is by definition equal to zero.

**Planned dose intensity (PDI)** is the assigned dose by unit of time planned to be given to patients as per protocol in the same dose unit and unit of time as that of the DI, i.e.

PDI (*dosing unit / unit of time*) = Planned cumulative dose (*dosing unit*) / Duration of exposure (*unit of time*).

For Part 2 of the study, note that only cyclosporine is administered and it is with a tapering regime.

For cyclosporine use 10 mg/kg/day as the planned dose for the first record and after that use the "prescribed dose x 2" as the planned dose and the "total daily dose" as the actual dose for exposure calculations. Summarise results in mg/kg/day.

For eltrombopag use 150 mg/day (or 100 mg/day for E/SE Asian patients) for planned dose for all records and "total daily dose" as the actual dose. Summarise results in mg/day.

Relative dose intensity (RDI) is defined as follows:

```
RDI = DI (dosing unit / unit of time) / PDI (dosing unit / unit of time).
```

```
e.g. RDI = DI (92.7 \text{ mg/day}) / PDI (100 \text{ mg/day}) = 0.927
```

### Study day

The study day describes the relative day of the event related to the start date of study treatment.

The reference start date is designated as **Study Day 1.** Study Day –1 is the day that precedes Day 1. Study Day 0 is not defined. Study day is not to be used in numerical computations, for example in calculating exposure.

The study day will be calculated as:

- The date of the event (visit date, onset date of an event, assessment date etc.) reference start date + 1, if event is on or after the reference start date.
- The date of the event (visit date, onset date of an event, assessment date etc.) reference start date, if event precedes the reference start date.

The reference start date for all assessments (safety, efficacy, patient reported outcomes (PROs), etc.) will be the start date of study treatment.

The study day will be displayed in the data listings. If an event starts before the reference start date, the study day displayed in the listing will be negative.

### **Baseline**

Baseline is the result of an investigation describing the "true" uninfluenced state of the patient, defined as the period from the date of signing any informed consent document to the start date of study treatment. Assessments, specified to be collected post-dose on the first date of study treatment are not considered.

The last non-missing assessment, including unscheduled assessments on or before the date of start of study treatment is defined as "baseline value" or "baseline assessment".

Where multiple measurements meet the baseline definition, with no further flag or label that can identify the chronological order, then values from central assessments should be considered as baseline rather than local values.

For electrocardiogram (ECG) parameters, if there are multiple replicates per time point, the average of these measurements would be calculated for baseline (if not already available in the database).

If patients have no value as defined above, the baseline result will be missing.

### Observation periods

The overall observation period will be divided into three mutually exclusive segments:

- 1. **Pre-treatment**: from day of patient's informed consent to start date of study treatment
- 2. **On-treatment**: from start date study treatment to last date of study treatment + 30 days
- 3. **Post-treatment**: from last date of study treatment + 31 days

#### On-treatment assessments/events

The definition of on-treatment is given below, depending on the context.

For safety summary tables an on-treatment AE is defined as any AE reported in the following time interval (including the lower and upper limits):

<date of first administration of study treatment; date of last administration of study treatment + 30 days>

This corresponds to the definition of treatment-emergent AEs given in the protocol, i.e. AEs which are newly reported or worsening from baseline.

An on-treatment assessment is defined as any assessment performed after the date of first administration of study treatment (except for assessments specified to be collected post-dose on that day), i.e. assessments performed in the following time interval (including the lower and upper limits):

• <date of first administration of study treatment + 1; date of last administration of study treatment + 30 days>

For patients whose last date of study treatment is missing, on-treatment assessments/events include any assessment/event present in the database occurring after the start date of study treatment.

Listings will contain all data, flagging assessments/events outside of the on-treatment period where applicable.

#### **Definition of Months and Years**

A month will be calculated as (365.25 / 12) = 30.4375 days. If duration is to be reported in months, duration in days will be divided by 30.4375. If duration is to be reported in years, duration in days will be divided by 365.25.

### Time since initial SAA diagnosis

Time since initial SAA diagnosis (days) = First dose date (Epag/CsA) – date of initial diagnosis.

### Time windows

Time windows for assessments are based on protocol specified windows. Weekly and biweekly visits should be completed  $\pm$  1 day. Biweekly visits after 6 months should be completed  $\pm$  2 days. Monthly visits should be completed  $\pm$  3 days. Bimonthly visits should be completed  $\pm$  1 week.

### Time windows for multiple assessments

In order to summarise data of assessments collected over time (including any unscheduled visits), the assessments will be time slotted. If more than one assessment is done within the same time window, the assessment performed closest to the target date will be used. If 2 assessments within a time window are equidistant from the target date, then the earlier of the 2 assessments will be used. If multiple assessments on the same date then the worst case will be used. The end of treatment assessment will be included if collected within 30 days of the last treatment date. Data from all assessments (scheduled and unscheduled), including multiple assessments, will be listed.

#### Last contact date

The last contact date will be derived for patients not known to have died at the analysis cut-off date using the latest complete date among the following:

Table 2-1 Last contact date data sources

| Source data | Conditions |
|---|---|
| Date of withdrawal of consent | Withdrawal of study informed consent |
| Date of discontinuation/phase completion | On the last disposition page completed |
| Start/End dates from drug administration records | Both study drugs. Doses of 0 are allowed |
| Sample collection dates | Sample collection marked as 'done' e.g. laboratory or pharmacokinetics (PK) |
| Assessment dates | At least one non-missing parameter value e.g. vital signs weight value, performance status available etc. |
| Start/End dates of AEs, medications or surgeries | Non-missing verbatim term |

The cut-off date will not be used for last contact date, unless the patient was last seen or contacted on that date. No date post cut-off date will be used. Completely imputed dates (e.g. the analysis cut-off date programmatically imputed to replace the missing end date of a dose administration record) will not be used to derive the last contact date.

The last contact date will be used for censoring of patients in the analysis of duration of hematological response.

### 2.2 Analysis sets

Patients who did not sign an informed consent form will be excluded from all analysis sets. All screened patients will be used in selected outputs.

### 2.2.1 Full Analysis Set

The Full Analysis Set (FAS) includes all patients who received at least one dose of study treatment (eltrombopag or cyclosporine).

### 2.2.2 Safety Set

The Safety Set includes all patients who received at least one dose of study treatment (eltrombopag or cyclosporine).

### 2.2.3 Per-Protocol Set

The Per-Protocol Set (PPS) includes the patients in the FAS who had no major protocol deviations.

The list of protocol deviations in Table 2-2 will lead to exclusion of the patient from the PPS.

Table 2-2 Protocol deviations leading to exclusion of patients from PPS

| PD description | Protocol deviation ID |
|---|---|
| Informed consent not obtained | INCL01 |
| SAA characterization not met | INCL03 |
| Evidence of clonal hematologic bone marrow disorder on cytogenetics* | EXCL02 |
| Prior immunosuppressive therapy with cyclosporine, alemtuzumab, rabbit or horse ATG and thrombopoietin receptor (TPO-R) agonists. | EXCL03 |
| Hypersensitivity to eltrombopag or its components | EXCL04 |
| Administration of an investigational drug within 30 days or 5 half-lives, whichever is longer, preceding the first dose of study treatment | EXCL11 |
| Eltrombopag starting dose not correct | TRT01 |
| Cyclosporine starting dose not correct | TRT02 |
| Failure to withdraw eltrombopag despite various reasons | WTH02 |
| Patient impacted by COVID19 | OTH02,-03,-04,-06 &<br>TRT10,-11 |

<sup>\*</sup>In addition the 4 patients who were enrolled and then discontinued from the study based on discrepancies between the local and central bone marrow assessment will be excluded – Using discontinued study with reason "Technical problems"

### 2.2.4 Pharmacokinetic Analysis Set

The Pharmacokinetic Analysis Set (PAS) includes all patients who provide at least one evaluable pharmacokinetics (PK) concentration. For a concentration to be evaluable, patients are required to:

- For samples on Week 2
  - take the same dose of eltrombopag for all dosing days prior to sampling on Week 2
  - for pre-dose sample, do not vomit within 4 hours after the dosing of eltrombopag prior to sampling
  - for post-dose samples, do not vomit within 4 hours after the dosing of eltrombopag on the sampling day
- For all pre-dose samples, have the sample collected before the next dose administration

### 2.2.5 Screening failures

Patients who sign an informed consent form but fail to start on study treatment for any reason will be considered a screen failure.

### 2.2.6 Subgroups of interest

The following subgroups of interest may be used in analyses:

- Age ( $<60, \ge 60 \text{ years}$ )
- Ethnicity (East/South East (E/SE) Asian vs Other)
- Responder status (Responder, Non-responder) see Section 2.5.1 for definition

# 2.3 Patient disposition, demographics and other baseline characteristics

The Full Analysis Set (FAS) will be used for all baseline and demographic summaries and listings unless otherwise specified.

### 2.3.1 Patient disposition

Disposition data will be summarised descriptively and listed. Summaries will include number and percentage (%) of patients who; complete a study phase (screening, treatment period 1, treatment period 2, post treatment follow-up and/or treatment discontinuation follow-up), patients who continue to the next phase, patients who discontinue a study phase with primary reason as reported on the disposition eCRF pages. Number (%) of patients who permanently discontinued study treatment with reason, as reported in the dose administration record eCRF pages will also be provided.

Informed consent and inclusion/exclusion criteria data will also be listed.

Data will be listed for screening failures.

The denominator will be based on the number of patients who enter the respective study phase (4 phases are used under PA1 and 2 phases are used under PA2, see study design figures in Section 1.1).

## 2.3.2 Patient demographics and other baseline characteristics

Demographic and other baseline data (e.g. medical history, transfusion history, diagnosis and extent of cancer, and eastern cooperative oncology group (ECOG) performance status etc.) will be summarised descriptively and listed. Age by category will also be summarised.

Demographic data for screen failure patients will be listed.

Demographic data will also be summarised by age sub-groups, ethnicity and/or responder status.

### **Medical history**

Medical histories and current medical conditions at baseline will be summarised separately for ongoing and historical medical conditions by primary system organ class (SOC) and preferred term (PT). Medical history and current medical conditions will be coded using the latest version of the Medical Dictionary for Regulatory Activities (MedDRA) at the time of analysis. Listings will be provided of all data.

### **Transfusion history**

Transfusion history for platelets and for red blood cells (RBCs) in the 4-weeks prior to initiation of dosing of eltrombopag and cyclosporine will be summarised and listed. The number of platelet/RBCs transfusions and time since last platelet/RBCs transfusion will be provided.

Time since last platelet/RBCs transfusion (in days) = Start date of treatment – start date of last platelet/RBCs transfusion.

### **Analyses sets**

The number (%) of patients in each analysis set (defined in Section 2.2) will be summarised.

# 2.4 Treatments (study treatment, concomitant therapies and compliance)

Eltrombopag (film-coated tablets) will be administered orally, once daily for 6 months. Cyclosporine (soft-gelatin capsules) will be administered orally, twice daily for the first 6 months and for a further 18 months (tapering regime for responder patients only). All patients must have safety evaluations for 30 days, after the last dose of study treatment.

### 2.4.1 Study treatment

Duration of study drug exposure (months), actual cumulative dose, actual dose intensity (DI) and relative dose intensity (RDI) will be summarised separately for each study drug (eltrombopag and cyclosporine) for the safety set.

The number of patients with dose changes, interruptions and permanent discontinuations will be presented, along with reasons for the dose change/interruption/permanent discontinuation for each study drug.

Duration of exposure (months) will also be categorized and summarised using the following time intervals:

- Eltrombopag:  $<1, \ge 1, \ge 2, \ge 3, \ge 4, \ge 5, \ge 6$
- Cyclosporine:  $<1, \ge 1, \ge 2, \ge 3, \ge 4, \ge 5, \ge 6, \ge 12, \ge 18, \ge 24$

Listings will be provided of all data.

### 2.4.2 Prior, concomitant and post therapies

Medications and significant non-drug therapies prior to and after the start of the study treatment will be coded according to the world health organization (WHO) Drug Reference List and summarised by anatomical therapeutic chemical (ATC) classification and preferred term.

Summary tables for concomitant medications and concomitant non-drug therapies for the safety set will be provided. Prior, concomitant and post study treatment medications and non-drug therapies will be listed for the safety set. Medications and therapies outside of the on-treatment period will be flagged.

Listings will be provided.

### 2.4.3 Protocol deviations

The number (%) of patients with protocol deviations will be summarised by deviation category (as specified in the latest version of the study data handling plan (DHP) at the time of analysis) and overall for the FAS. All protocol deviations will be listed, flagging those leading to the exclusion of a patient from an analysis set. Protocol deviations will be listed for screening failures (if any).

### 2.4.4 Handling of missing values

For analyses prior to the final analysis (at 24 months), if the date of last administration of study drug is completely missing and there is no end of treatment eCRF page, the patient is considered as on-going and the earliest of; death date, last contact date or cut-off date, will be used as the 'last dosing date' for calculation/derivation purposes e.g. durations. Last administration date should not be missing for the final analyses.

### 2.5 Analysis of the primary objective

The primary objective of this study is to evaluate the efficacy of eltrombopag+cyclosporine as first-line therapy as measured by the overall hematologic response rate by 6 months. That is, after all enrolled patients have completed 6 months of study treatment or discontinued study treatment or study prior to 6 months. Efficacy analyses and listings are based on the FAS.

# 2.5.1 Primary endpoint

The overall hematologic response rate (ORR) is defined as the proportion of patients achieving complete response (CR) and partial response (PR) defined as follows:

**Partial response** (PR) is defined as any two of the following parameters at two consecutive, scheduled visit measurements at least 7 days apart during the first 6 months of study (and not sufficient for CR) and no platelet transfusions within 7 days of platelet measurement (can still be a PR if ANC and reticulocyte measurements are valid):

- Absolute neutrophil count (ANC)  $\geq 500/\mu L$
- Platelet count  $\geq 20~000/\mu L$
- Reticulocyte count  $\geq 60~000/\mu L$  (automated)

Complete response (CR) is defined as all three parameters meet the following criteria at two consecutive, scheduled visit measurements at least 7 days apart during the first 6 months of study and no platelet transfusions within 7 days of platelet measurement and no RBC transfusion with 14 days of the hemoglobin measurements:

- ANC  $\geq 1~000/\mu L$
- Platelet count  $\geq 100 \ 000/\mu L$
- Hemoglobin  $\geq 10 \text{ g/dL}$

ORR\_6 = Number of patients who achieved hematologic response by 6 months/Number of patients in the FAS.

**Responder status**: If any patient achieves hematologic response (either CR or PR) any time on or before the 6 months visit, they will be considered a **responder**, else they are a **non-responder**.

The point estimate along with the corresponding exact 95% confidence interval using Clopper and Pearson exact method will be presented for ORR 6.

Day 10 (plat 8 000) sample at 10:00 and platelet transfusion Day 10 11:00 (plat 60 000)— assume transfusion is always after the blood sample Day 10 sample is valid for efficacy.

Day 11 to Day 16 not valid (Day 11 (50 000), 12 (45 000), 13, 14, 15, 16 (transfusion minimal impact by day 7) not valid). Both Day 10 and Day 17 samples are valid for efficacy

### Handling of missing values/discontinuations

If any patient achieves overall hematologic response any time before 6 months but discontinues prior to 6 months or has missing parameters required for assessing overall hematologic response at any point after achieving the first response, they will be considered as responders.

Due to COVID19 situation some patients may have local instead of central lab results for scheduled visits. For all patients, local results (including the visit window period) will be used if all 4 results of the efficacy parameters (hemoglobin, neutrophils, reticulocytes, platelets) from the central laboratory are not available for a scheduled visit.

### 2.5.2 Supportive analyses

The ORR by 6 months (primary analysis) will be repeated on the PPS.

The ORR by 6 months (primary analysis) will also be summarised by age sub-groups and/or ethnicity using the FAS and/or PPS.

The ORR at 6 months will be summarised using the FAS as follows:

- The overall hematologic response will be calculated at 6 months (based on assessment at 6 months visit and the previous visit at least 7 days apart) based on the evaluable patients (i.e., patients for whom data is available at 6 months). Thus if a patient has missing laboratory parameters at 6 months or the prior visit at least 7 days apart required to calculate CR or PR, or if the patient discontinued earlier than 6 months, then the patient will be considered as a non-responder.
- ORR\_a6 = Number of patients who achieved hematologic response at 6 months/Number of patients in the FAS.

## 2.6 Analysis of secondary efficacy objective(s)

All secondary efficacy analyses will be performed on the FAS, unless otherwise specified.

Secondary objectives will be summarised in the 6 and 24 months CSRs with data reported cumulatively. Listings will be provided.

### 2.6.1 ORR by 3 months, at 12 months and at 24 months

The ORR by 3 months will be evaluated and summarised as for the ORR by 6 months, i.e. if any patient achieves hematologic response any time on or before the month 3 visit, they will be considered a **3 month responder**, else they are a **3 month non-responder**.

- ORR\_3 = Number of patients who achieved hematologic response by 3 months/Number of patients in the FAS.
- The ORR by 3 months will be repeated on the PPS.
- The ORR **by** 3 months will also be summarised by age sub-groups and/or ethnicity using the FAS and/or PPS.

The ORR at 12 months and at 24 months will be summarised as for the ORR at 6 months. If any 6 month responder achieves hematologic response at 12 months (24 months) visit, they will be considered at **12 months** (24 months) **responder**, else they are at **12 month** (24 month) **non-**

**responder**. The 12 months (24 months) visit will be the confirmatory visit of the most recent visit assessment prior to this assessment (at least 7 days apart).

- ORR\_a12 (ORR\_a24) = Number of patients who achieved hematologic response at 12 months (24 months)/Number of patients in the FAS.
- The ORR at 12 months (24 months) will be repeated on the PPS.
- The ORR at 12 months (24 months) will also be summarised by age sub-groups and/or ethnicity using the FAS and/or PPS.

### 2.6.2 Duration of hematologic response

The time from start of the first hematologic response (the initial assessment, not the confirmatory assessment, of either CR or PR whichever occurs first by 6 months) to the date of first relapse will be derived as:

• Duration of first hematologic response (days) = End date (Date of first relapse) – start date of first hematologic response + 1

Longest duration will also be presented:

• Longest duration of hematologic response (days) = End date (Date of relapse) – start date of longest hematologic response + 1

**Relapse** is defined as no longer meeting the definition of PR (and not CR).

The duration of hematological response will be estimated using Kaplan-Meier method and the median time to relapse will be presented along with 95% confidence interval. If no relapse occurs, the patient will be **censored** at the date of last contact.

### 2.6.3 Relapse rate

The number (%) of responders who relapse during the study will be reported by 6 and 24 months on a cumulative basis and will be summarised together with the corresponding exact 95% confidence interval using Clopper and Pearson exact method.

### 2.6.4 Clonal evolution

The number (%) of patients along with corresponding exact 95% confidence interval (using Clopper and Pearson exact method) with possible clonal evolution to myelodysplasia, paroxysmal nocturnal hemoglobinuria (PNH) and/or acute leukemia occurring during the study will be summarised by 6 and 24 months. Clonal evolution to each group is defined as:

- **myelodysplasia**: a new marrow cytogenic abnormality with complex karyotype marked as 'Yes'
  - taken from the 'Cytogenetics / Other Abnormalities' eCRF page.
- PNH: a clone of peripheral blood GPI-deficient (%) having cumulative PNH sub-type of type 2 RBC% and type 3 RBC% value of <10% at baseline that rose to >50% on study
  - taken from the 'Flow cytometry' eCRF page using the parameter 'Peripheral blood GPI-deficient (%)'
  - Any rise (local or central) will be considered
- acute leukemia: >20% peripheral blood and/or marrow blasts post baseline

• marrow blasts are taken from the 'Bone Marrow Aspirate' or the 'Bone Marrow Biopsy' eCRF page using the 'Blast Cells (%)' parameter

Programmed listing results will be reviewed by clinical and/or steering committee members and confirmed cases of clonal evolution will be discussed in the CSR.

### 2.6.5 Blood (RBC) and platelet transfusions

The number (%) of patients with corresponding 95% confidence interval (using Clopper and Pearson exact method) will be summarised by 6 and 24 months (responders only) for patients:

- who received at least one platelet transfusion
- who received at least one RBC transfusion
- with platelet transfusion independence
- with RBC transfusion independence

Transfusion independency is considered if transfusions are not required in at least a 28 day period for platelet transfusions and at least 56 day period for RBC transfusions.

In addition the duration of the longest interval without a platelet or RBC transfusion by 6 months and by 24 months (responders only) will be summarised using Kaplan-Meier analysis and the median longest duration will be presented along with 95% confidence interval.

- Longest duration of platelet transfusion independence (days) = End date of longest interval start date of longest interval + 1
- Longest duration of RBC transfusion independence (days) = End date of longest interval start date of longest interval + 1

### Note that:

- the start date of the longest interval might use the patient's first dose date or the patient's last transfusion date + 1
- the end date of the longest interval might use the patient's first transfusion date 1 or if no end date of longest interval without a platelet or RBC transfusion occurs, the patient will be **censored** at the date of last contact.

Listings will be provided.

Transfusions packed red blood cells, platelets and longest duration of transfusion independence will be also summarised by age sub-groups and/or ethnicity.

### 2.7 Safety analyses

Safety analyses will be based on the safety set unless otherwise specified. The summary tables will be presented for 'Responders', 'Non-responders' and 'All subjects' where indicated. Listings will be provided.

## 2.7.1 Adverse events (AEs)

The AEs will be coded using the latest version of MedDRA at the time of the analysis. AEs will be graded using the common toxicity criteria for adverse events (CTCAE) Version 4.03

AE summaries will only include AEs during the on-treatment period. A column for 'Grade  $\geq$  3' may be included in the AE tables. If a patient reported more than one AE with the same preferred term (PT), the AE with the greatest severity will be presented. If a patient reported more than one AE within the same primary system organ class (SOC), the patient will be counted only once with the greatest severity at the SOC level, where applicable. An AE with missing CTCAE grade will be included in the 'All grades' column of the summary tables.

In AE summaries, the primary SOC will be presented alphabetically and the PTs will be sorted within the primary SOC in descending frequency.

Summary tables will be provided for:

- Overview of AEs
  - In-text table
- All AEs regardless of relationship to study treatment by primary SOC, PT and maximum severity and age as well as ethnicity
  - In-text table by SOC and maximum severity
  - In-text table by PT and maximum severity
- AEs suspected to be related to study treatment by SOC, PT and maximum severity
  - In-text table by PT and maximum severity
- AEs leading to study treatment discontinuation regardless of relationship to study treatment by SOC, PT and maximum severity
  - In-text table by PT and maximum severity
- AEs leading to study treatment discontinuation suspected to be related to study treatment by SOC, PT and maximum severity
- AEs leading to study treatment adjustment and/or interruption regardless of relationship to study treatment by SOC, PT and maximum severity
- SAEs regardless of relationship to study treatment by SOC, PT and maximum severity
  - In-text table by PT and maximum severity
- SAEs suspected to be related to study treatment by SOC, PT and maximum severity
- On-treatment deaths and SAEs suspected to be related to study treatment by SOC and PT
- Non-SAEs regardless of relationship to study treatment (threshold 0-5%) by SOC and PT
- On-treatment deaths by SOC and PT and age, ethnicity as well as responder status
  - In-text table by SOC and PT
- All deaths by SOC and PT and responder status

All AEs will be listed. AEs outside of the on-treatment period will be flagged.

# Adverse events of special interest / grouping of AEs

The adverse events of special interest (AESI) are maintained and updated on a regular basis in the project case retrieval sheet (CRS) and the latest version at the time of the analyses will be used. An in-text and post-text summary table by SOC, PT and maximum severity will be provided.

An AESI is a grouping of AEs that are of scientific and medical concern specific to eltrombopag. These groupings are defined using MedDRA terms, standardized MedDRA queries (SMQs), high level group terms (HLGTs), HLT (high level terms) and PTs. Customized SMQs called Novartis MedDRA queries (NMQs) may also be used. A NMQ is a customized group of search terms which defines a medical concept for which there is no official SMQ available or the available SMQ does not completely fit the need. It may include a combination of single terms and/or an existing SMQ, narrow or broad. For each specified AESI, number (%) of patients with at least one event of the AESI occurring during on-treatment period will be summarised by responder status and overall.

A listing of AESIs will be provided and a listing of all grouping levels down to the MedDRA preferred terms used to define each AESI will be generated.

### **2.7.2** Deaths

See Section 2.7.1. A listing will be provided of all deaths, deaths outside of on-treatment period will be flagged. This all deaths listing will be for "All screened patients" so that deaths during screening are also presented.

### 2.7.3 Laboratory data

Laboratory values (central and local) are converted to the international system of units (SI). CTCAE Grade 0 will be assigned for all non-missing values not graded as 1 or higher. Grade 5 will not be used. For laboratory tests where grades are not defined by CTCAE version 4.03, results will be categorized as low/normal/high based on laboratory normal ranges.

The following summaries will be generated separately for hematology and for the safety set:

- Shift tables by CTCAE grade (or low/normal/high classification) to compare baseline to the worst on-treatment value:
  - Hematology: Neutrophils (absolute), platelets and hemoglobin
  - Chemistry: Creatinine, total bilirubin (TBL), aspartate aminotransferase (AST), alanine aminotransferase (ALT) and alkaline phosphatase (ALP)
- Summary statistics on platelets for change from baseline for months 3, 6, 12 and 24 will be provided. On-treatment platelet values will be used up to Month 24.
- Box plots showing parameter values over time (baseline and on-treatment time points 3, 6, 12 and 24 months) will be displayed based on time windows for the following selected parameters: Neutrophils (absolute), platelets, reticulocytes, hemoglobin and RBCs. Boxplots will display boxes (25<sup>th</sup> 75<sup>th</sup> percentiles) and median (line) as well as joint mean (dot) values. Whiskers extend to the 10<sup>th</sup> 90<sup>th</sup> percentiles with any values outside the whiskers not being displayed. A footnote will explain that these values are not displayed. However, all values are used to calculate mean and percentiles displayed on the graph. The number of observations used for this analysis is to be stated at the bottom.

Listings of laboratory data (hematology and biochemistry) will be provided showing the corresponding CTCAE grades, if applicable, and the classifications relative to the laboratory normal ranges. Values measured outside of on-treatment period will be flagged.

### Liver function parameters

Liver function parameters of interest are TBL, ALT, AST and ALP.

The number (%) of patients with worst on-treatment values will be summarised:

- ALT or AST > 3xULN
- ALT or AST > 5xULN
- ALT or AST > 8xULN
- ALT or AST > 10xULN
- ALT or AST > 20xULN
- TBL > 2xULN
- TBL > 3xULN
- ALT or AST > 3xULN & TBL > 2xULN
- ALT or AST  $> 3xULN \& TBL > 2xULN \& ALP \ge 2xULN$
- ALT or AST > 3xULN & TBL > 2xULN & ALP < 2xULN (potential Hy's law)

Listings of liver event data will be provided. Values measured outside of on-treatment period will be flagged.

### 2.7.4 Other safety data

### 2.7.4.1 ECG

12-lead ECGs, including QTcF (Fridericia's correction), mean heart rate (HR), PR-, QT- and QRS-durations, will be obtained locally for each patient during the study. ECG data will be read and interpreted locally.

Where ECG replicates are provided for an assessment, the average of the ECG parameters at that assessment will be used in the analyses.

The number (%) of patients with notable values will be presented.

Table 2-3 Notable criteria for ECG parameters

| Parameter | Notable low value | Notable high value |
|---|---|---|
| QTcF | | New value of >450 and ≤ 480 ms New value of >480 and ≤ 500 ms New value of >500 ms Increase from baseline of >30 ms to ≤ 60 ms Increase from baseline of >60 ms |
| Heart rate | Decrease >25% from baseline and to a value <50 bpm | Increase >25% from baseline and to a value >100 bpm |
| PR | | Increase >25% from baseline and to a value >200 ms<br>New value of >200 ms |
| QRS | | Increase >25% from baseline and to a value >120 ms New value of >120 ms |

A listing of all ECG assessments will be produced. Notable values as well as values measured outside of on-treatment period will be flagged in the listings.

### 2.7.4.2 Vital signs

Vital sign assessments are performed in order to characterise basic body function. The following parameters were collected: height (cm, inch), weight (kg, pound), body temperature (°C, Fahrenheit), position, pulse (beats/minute), systolic and diastolic blood pressure (mmHg).

The number (%) of patients with notable values will be presented.

Table 2-4 Notable criteria for vital signs

| Vital sign (unit) | Notable low value | Notable high value |
|---|---|---|
| Weight (kg) | decrease ≥ 10% from baseline | increase ≥ 10% from baseline |
| Body temperature (°C) | | ≥ 39.1 |
| Pulse rate (bpm) | ≤ 50 and decrease from baseline of >25% | ≥ 100 and increase from baseline of >25% |
| Systolic blood pressure (mmHg) | ≤ 90 and<br>decrease from baseline of ≥ 20 | ≥ 180 and<br>increase from baseline of ≥ 20 |
| Diastolic blood pressure (mmHg) | ≤ 50 and<br>decrease from baseline of ≥ 15 | ≥ 105 and increase from baseline of ≥ 15 |

A listing of all vital sign assessments will be produced and notable values will be flagged. Assessments collected outside of on-treatment period will be flagged.

### **ECOG** performance status

The eastern cooperative oncology group (ECOG) performance status will be used to assess physical health of patients, ranging from 0 (most active) to 5 (least active).

Shift tables comparing the baseline status with the worst post-baseline status will be provided.

Table 2-5 ECOG performance scale

| Score | Description |
|---|---|
| 0 | Fully active, able to carry on all pre-disease performance without restriction |
| 1 | Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work |
| 2 | Ambulatory and capable of all self-care but unable to carry out any work activities. Up and about more than 50% of waking hours |
| 3 | Capable of only limited self-care, confined to bed or chair more than 50% of waking hours |
| 4 | Completely disabled. Cannot carry on any self-care. Totally confined to bed or chair |
| 5 | Dead |

A listing of all ECOG performance status assessments will be produced, flagging assessments collected outside of the on-treatment period.

### Ophthalmic and neurologic examinations

No summaries or listings as only collected as source data.

### 2.8 Pharmacokinetic endpoints

The PAS will be used for the PK data analysis and the FAS for the listings.

PK parameters for eltrombopag will be determined using non-compartmental methods using Phoenix (Pharsight, Mountain View, CA) or other appropriate software. PK parameters listed in the table below will be estimated and reported, when feasible.

Table 2-6 Non-compartmental PK parameters of eltrombopag

| Parameter | Description |
|---|---|
| Cmax | Observed maximum plasma concentration following administration (mass/volume) |
| AUClast | Area under the curve calculated to the last quantifiable concentration point (Tlast) (mass*time/volume) |
| AUCtau | Area under the curve calculated to the end of the dosing interval (tau) (mass*time/volume) |
| Ctrough | Pre-dose plasma concentration (mass/volume) |
| Tmax | The time to reach peak or maximum concentration (time) |
| CLss/F | Apparent systemic (or total body) clearance at steady state from plasma (volume/time) |

The concentrations obtained for the Week 2 pre-dose sample (sample 1) will be duplicated in order to also be analysed as a 24 h post-dose sample (and will be attributed sample number 6 for analysis purposes).

Descriptive statistics of all PK parameters and PK concentrations will include arithmetic and geometric mean, median, sd, and coefficient of variation (CV), geometric CV, minimum and maximum. Zero concentrations will not be included in the geometric mean calculation. Since Tmax is generally evaluated by a nonparametric method, only n, median values and ranges will be given for this parameter.

PK parameters and PK concentrations will be summarized descriptively by ethnicity subgroups (if at least 3 patients with PK parameters and/or concentrations in the subgroup) and overall. The PK parameters, Cmax, AUClast, AUCtau, and Ctrough, will be normalized to the protocol starting dose i.e. 100 mg for S/SE Asians and 150 mg for Others.

Individual PK concentrations will be listed. The PK sample/concentrations will be flagged in the listing when:

- 1- Patient changed or interrupted the dose during 7 days before PK sample collection
- 2- Patient changed the dose during the 2 weeks before PK sample collection
- 3- Patient vomited within 4 hours after dosing on day of PK assessment for post-dose samples, or on the day prior to sampling, for pre-dose samples
- 4- PK sample was collected out of time interval for the 24-hour sample, the time window considered is 20-28 hours

These flags will be programmatically set up during the PK merge with the clinical database. For the first three PK flags the sample will be excluded from the analysis for PK parameter calculation and from the descriptive statistics of concentrations over scheduled sample

collection time. For the fourth PK flag the sample will be excluded from the descriptive statistics of concentrations over scheduled sample collection time only.

In addition, during analysis the pharmacokinetics will flag PK samples/concentrations when dose, sample collection time and/or concentration value are missing, as well if pre-dose samples are collected post-dose. Those PK samples/concentrations will be excluded from the analysis for PK parameter calculation and from the descriptive statistics of concentrations over scheduled sample collection time.

All individual PK parameters and PK concentrations will be listed. Those PK concentrations or PK parameters not evaluable for statistical analysis will be flagged and the reason for exclusion will be given in the listings.

The following analyses and results may be performed and reported separately from the CSR:

Exposure-response analysis will be conducted, if supported by the data to evaluate relationship between exposure of eltrombopag and response and specific AEs of special interests. These relationships will be explored by graphical methods. Any apparent relationship may be further characterized by a model as appropriate and supported by the data.

Population PK may be performed if supported by the data to explore relevant covariates.

### Handling of PK data below LLOQ or missing

Missing concentration values will be reported as such in data listings. Concentration values below the LLOQ will be handled as zero in summary statistics, and reported as such in data listings. Any missing PK parameter data will not be imputed.

# 2.9 Patient-reported outcomes (PROs)

The FAS will be used for analysing PRO data unless otherwise specified. The summary tables will be presented for 'Responders', 'Non-responders' and 'All subjects'. Listings will be provided. Box plots showing parameter values over time will be displayed, as applicable. Boxplots will display boxes  $(25^{th} - 75^{th})$  percentiles) and median (line) as well as joint mean (dot) values. Whiskers extend to the  $10^{th} - 90^{th}$  percentiles with any values outside the whiskers not being displayed.

# 2.9.1 FACIT-Fatigue and FACT-TH18 (includes FACT-G)

Functional assessment of chronic illness therapy (FACIT)-Fatigue, functional assessment of cancer therapy-thrombocytopenia 18 (FACT-TH18) and functional assessment of cancer therapy-general (FACT-G) responses will be generated in accordance with the respective scoring manual. Descriptive statistics will be used to summarise the actual subtotal/total score and absolute change from baseline to each visit assessment. Patients with an evaluable baseline score and at least one evaluable post baseline subtotal/total score during the on-treatment period will be included in the change from baseline analyses.

Missing responses for items in a scale will be handled based on the respective instrument manual. All PRO analyses will include data as imputed according to the scoring manual. No imputation will be applied if the total or subscale scores are missing at a visit.

### **FACIT-Fatigue**

There are 13 items. Negatively worded items are reverse scored prior to summing. Add the scores together, multiply by 13 and then divide by the number of items answered. A total score of <30 indicates severe fatigue. The higher the total score the better the quality of life. Total score can vary from 0 to 52.

In cases some answers are missing, a total score is prorated from the score of the answered items, so long as more than 50% of the items (i.e., at least 7 of 13) were answered.

Further details on the **FACIT-Fatigue** scoring is provided in Appendix 6.4 and at:

http://www.facit.org/FACITOrg/Questionnaires

http://www.physio-pedia.com/Functional\_Assessment\_of\_Chronic\_Illness\_Therapy

#### **FACT-TH18 and FACT-G**

There are 27-items divided into 4 domains in the FACT-G part, Physical Well-Being (PWB), Social/Family Well-Being (SWB), Emotional Well-Being (EWB), Functional Well-Being (FWB). Calculate the total scores for each subscale and overall in a similar way as for the FACIT-Fatigue, i.e. after reversing the scoring of negatively worded items (so that a higher score always indicated a favorable response), item responses are summed.

In cases where some answers may be missing, a total score is prorated from the score of the answered items, so long as more than 50% of the items were answered. E.g. for PWB, where PWB\_N = N(OF GP1-GP7) i.e. number of items not missing in GP1 to GP7

IF (PWB N/7 > 0.50) THEN PWB = SUM(OF GP1-GP7) \*7/(PWB N);

Note that a total score should only be calculated if ALL of the component subscales have valid scores.

Summary of the total scores:

- FACT-G total score: PWB score + SWB score + EWB score + FWB score
- FACT-Th total score: PWB score + SWB score + EWB score + FWB score + ThS score i.e. FACT-Th total score = FACT-G total score + Th subscale score
- FACT-Th Trial Outcome Index (TOI): PWB score + FWB score + ThS score

Further details on FACT-TH18 and FACT-G scoring is provided in Appendix 6.4 and at:

https://www.rtog.org/LinkClick.aspx?fileticket=bAZw9mE3jlQ%3D&tabid=118

For business use only

Novartis





# 2.11 Interim analysis

There are 2 planned reporting events, each with a CSR:

- Primary analysis (6 months)
- Final analysis (24 months)

# 3 Sample size calculation

50 patients will be enrolled in the study.

With 50 patients criteria

- a: observed overall hematologic response rate (ORR) ≥ "clinically meaningful" threshold (30%) and
- b: probability of true overall hematologic response rate "not being clinically meaningful (response ≤ 20%)" is less than 10%

will be met if at least 15 responders out of 50 patients treated with combination therapy, eltrombopag+cyclosporine are observed by 6 months.

With 54 patients the criteria will be met if at least 17 responders out of 54 patients are observed.

Table 3-1 Table showing observed response rate and its posterior distribution using a Beta-binomial model

| Sample size | No. of responders | Observed response rate (%) | Probability of 'not being clinically meaningful (response rate ≤20%)" |
|---|---|---|---|
| N=50 | 13 | 26.0 | 0.1693 |
| | 14 | 28.0 | 0.0992 |
| | 15 | 30.0 | 0.0538 |
| | 16 | 32.0 | 0.0269 |
| | 17 | 34.0 | 0.0125 |
| N=54 | 14 | 25.9 | 0.1618 |
| | 15 | 27.8 | 0.0961 |
| | 16 | 29.6 | 0.0530 |
| | 17 | 31.5 | 0.0272 |
| | 18 | 33.3 | 0.0130 |

For example, if 15 responders out of 50 patients are observed, the observed ORR will be 30% and the posterior probability that  $\theta \le 20\%$  is 0.0538. The latter is found using the posterior distribution  $\theta | Y \sim \text{Beta}(0.25 + 15, 1 + 50 - 15)$ . In R this would be calculated as pbeta (0.2, 15.25, 36).

The operating characteristics of the design are presented in the table below. This table shows the probability of a positive conclusion (i.e. success criteria met at the end of the study) under different underlying true response rates. When the effect of the combination therapy is not clinically meaningful (true response rate  $\leq 20\%$ ), the probability of a positive conclusion is <10% (false success rate). The probability of success is >94% when the true response rate by 6 months is 40%.

| Table 3-2 Operating characteristics of the study | / design |
|--------------------------------------------------|----------|
|--------------------------------------------------|----------|

| Sample size | True response rate (%) | Probability of positive conclusion |
|-------------|------------------------|------------------------------------|
| N=50 | 10 | 0.0001 |
| | 20 | 0.0607 |
| | 30 | 0.5532 |
| | 40 | 0.9460 |
| | 50 | 0.9987 |
| N=54 | 10 | 0.0000 |
| | 20 | 0.0310 |
| | 30 | 0.4567 |
| | 40 | 0.9235 |
| | 50 | 0.9981 |

From Table 3-1 it is known that at least 15 responders need to be observed in 50 patients for study success. The operating characteristics in Table 3-2 are now the probabilities under a given assumed true ORR to observe  $\geq 15$  responders. For example, if the assumed true response rate is 40%, this probability is 0.9460 and is found by using the cumulative binomial distribution function. In R, this would be calculated as 1 - pbinom (14, 50, 0.4).

## 3.1.1 Bayesian calculus for a binary endpoint

For the binary endpoint ORR, let Y be the number of responders in n subjects. The sampling model is binomial

$$Y \mid \theta \sim Bin(n, \theta)$$

with true response rate  $\theta$ . The prior distribution is a Beta distribution

$$\theta \sim Beta(a, b)$$

In this conjugate setting, the posterior distribution is again a Beta distribution

$$\theta \mid Y \sim Beta(a+Y, b+n-Y)$$

Here, the parameters a and b are the a priori number of responders and non-responders, respectively, and a+b is the prior effective sample size.

For this study, the parameters (a, b) of the Beta prior distribution are a = 0.25 and b = 1. This prior distribution has mean = a / (a + b) = 0.25 / (0.25 + 1) = 0.2 assuming a low response rate a priori. Furthermore, the prior effective sample size is small (a + b = 1.25).

# 4 Changes to protocol specified analyses

Supportive efficacy analyses were added as specified in Section 2.5.2.

Not all laboratory and liver event data will be listed, listings for key biochemistry, hematology and hepatic parameters will be provided.

Sample size characteristics were added based on the enrollment of 54 patients.

Age categories is changed to <60, >=60. Additional subgroups analysis by age, ethnicity and/or responder status were added for demographic characteristics, overall hematological response, transfusion information and relevant AEs.

Boxplots displaying parameter values over time for the patient-reported outcomes were added.

### 5 References

- 1. Brookmeyer R and Crowley J (1982). A Confidence Interval for the Median Survival Time. Biometrics, 38, 29 41.
- 2. Clopper CJ and Pearson ES (1934). The use of confidence or fiducial limits illustrated in the case of the binomial. Biometrical, 26, 404-413.
- 3. Collet D (1994). Modelling survival data in medical research. London, Chapman & Hall.
- 5. Neuenschwander B, Branson M and Gsponer T (2008). Critical aspects of the Bayesian approach to Phase I cancer trials. Statistics in Medicine, 27, 2420-2439.
- 6. Oncology guideline for safety analysis, v1.0, dated 09-Jun-2016
- 7. Spiegelhalter DJ, Abrams KR and Myles JP (2004). Bayesian Approaches to Clinical Trials and Health-care Evaluation. Chichester, Wiley.

# 6 Appendix 1

# 6.1 Imputation rules

# 6.1.1 AE, concomitant medication (CM) and safety assessment date imputation

Table 5-1 Imputation of start dates (AE, CM) and assessments (LB, EG, VS)

| Missing<br>Element | Rule |
|---|---|
| day, month, and year | No imputation will be done for completely missing dates |
| day, month | <ul> <li>If available year = year of study treatment start date then <ul> <li>If stop date contains a full date and stop date is earlier than study treatment start date then set start date = 01JanYYYY</li> <li>Else set start date = study treatment start date.</li> </ul> </li> <li>If available year &gt; year of study treatment start date then 01JanYYYY</li> <li>If available year &lt; year of study treatment start date then 01JulYYYY</li> </ul> |
| day | <ul> <li>If available month and year = month and year of study treatment start date then <ul> <li>If stop date contains a full date and stop date is earlier than study treatment start date then set start date= 01MONYYYY.</li> <li>Else set start date = study treatment start date.</li> </ul> </li> <li>If available month and year &gt; month and year of study treatment start date then 01MONYYYY</li> <li>If available month and year &lt; month year of study treatment start date then 15MONYYYY</li> </ul> |
| LB: Laborator | ry, EG: ECG, VS: Vital signs |

Table 5-2 Imputation of end dates (AE, CM)

| Missing<br>Element | Rule (*=last treatment date plus 30 days not > (death date, cut-off date, withdrawal of consent date)) |
|---|---|
| day, month,<br>and year | Completely missing end dates (incl. ongoing events) will be imputed by the end date of the on-treatment period* |
| day, month | • If partial end date contains year only, set end date = earliest of 31DecYYYY or end date of the on-treatment period * |
| day | • If partial end date contains month and year, set end date = earliest of last day of the month or end date of the on-treatment period* |

Any AEs and CMs with partial/missing dates will be displayed as such in the data listings. Any AEs and CMs which are continuing as per data cut-off will be shown as 'ongoing' rather than the end date provided.

### 6.1.2 Prior therapies date imputation

Missing day is defaulted to the 15<sup>th</sup> of the month and missing month and day is defaulted to 01-Jan.

# 6.2 Laboratory parameters derivations

CTCAE grading for blood differentials is based on absolute values. However, this data may not be reported as absolute counts but rather as percentage of WBC.

If laboratory values are provided as '<X' (i.e. below limit of detection) or '>X', prior to conversion of laboratory values to SI unit, these numeric values are set to X.

The following rules will be applied to derive the WBC differential counts when only percentages are available for a xxx differential

```
xxx count = (WBC count) * (xxx %value / 100)
```

Further derivation of laboratory parameters might be required for CTCAE grading. For instance, corrected calcium can be derived using the reported total calcium value and albumin at the same assessment using the following formula:

Corrected Calcium (mg/dL) = Calcium (mg/dL) - 0.8 [Albumin (g/dL)-4]

In order to apply the above formula, albumin values in g/L will be converted to g/dL by multiplying by 0.1), calcium values in mmol/L will be converted to mg/dL by dividing by 0.2495. For calculation of laboratory CTCAE grades 0 and 1, the normal range for derived corrected calcium is set to the same limits (in mg/dL) as for calcium.

### 6.3 Statistical models

### 6.3.1 Primary analysis

### Calculation of posterior probability

The efficacy criteria for this study are:

- 1. Observed overall hematologic response rate ≥ "clinically meaningful" threshold (30%)
- 2. Probability of true overall hematologic response rate "not being clinically meaningful (response \le 20\%)" is less than 10\%

Let p denote the proportion of patients who achieves overall hematologic response by 6 months and follow a beta prior distribution Beta [a, b], where a>0, b>0. Let y out of n patients achieve overall hematologic response by 6 months. Therefore, the posterior distribution of p is Beta[a+y, b+ n-y] [Spiegelhalter et al. 2004].

A minimally informative unimodal Beta prior [Neuenschwander et al. 2008] Beta [0.25, 1] will be used. The parameters were chosen so that the posterior probability of the true response rate  $\leq 20\%$  (considered not clinically meaningful) is equal to 0.0538.

The efficacy criteria will be assessed based on the actual number of patients enrolled in the study. For example, if the total number of patients is 50, the efficacy criteria requires that at least 15 patients achieve overall hematologic response by 6 months. In that case, the posterior

distribution is Beta[0.25+15, 1+50-15] i.e. Beta[15.25, 36] and the probability of success is >90% when the true responder rate is 40%.

### Confidence interval for response rate

Responses will be summarised in terms of percentage rates with  $100(1 - \alpha)\%$  confidence interval using exact binomial confidence interval (implemented using SAS procedure FREQ with EXACT statement for one-way table [Clopper and Pearson 1934].

### 6.3.2 Key secondary analysis

### Kaplan-Meier estimates

An estimate of the survival function (i.e., time to relapse, duration of transfusion independence) will be constructed using Kaplan-Meier (product-limit) method as implemented in PROC LIFETEST with METHOD=KM option. The PROC LIFETEST statement will use the option CONFTYPE=LOGLOG.

Median survival will be obtained along with 95% confidence intervals calculated from PROC LIFETEST output using the method of [Brookmeyer and Crowley 1982]. Kaplan-Meier estimates of the survival function with 95% confidence intervals at specific time points will be summarised. The standard error of the Kaplan-Meier estimate will be calculated using Greenwood's formula [Collett 1994].

## 6.4 FACIT-Fatigue scoring guideline

FACIT-Fatigue Subscale Scoring Guidelines (Version 4) – Page 1

Instructions:\*

- 1. Record answers in "item response" column. If missing, mark with an X
- 2. Perform reversals as indicated, and sum individual items to obtain a score.
- 3. Multiply the sum of the item scores by the number of items in the subscale, then divide by the number of items answered. This produces the subscale score.
- 4. The higher the score, the better the OOL.

| <b>Subscale</b> | <b>Item Code</b> | Reverse iter | <u>n?</u> | <u>Item response</u> | <b>Item Score</b> |
|---|---|---|---|---|---|
| FATIGUE | HI7 | 4 | - | | = |
| SUBSCALE | HI12 | 4 | - | | = |
| | Anl | 4 | - | | = |
| | An2 | 4 | - | | = |
| Score range: 0-52 | An3 | 4 | - | | = |
| score range. 0 32 | An4 | 4 | - | | = |
| | An5 | 0 | + | | = |
| | An7 | 0 | + | | = |
| | An8 | 4 | - | | = |
| | An12 | 4 | - | | = |
| | An14 | 4 | - | | = |
| | An15 | 4 | - | | = |
| | An16 | 4 | - | | = |

Sum individual item scores:

| Multiply by 13: | |
|-------------------------------------|------------------|
| Divide by number of items answered: | = <u>Fatigue</u> |

### Subscale score

#### FACT-Th18 and FACT-G scoring guideline 6.5

**Scoring Guidelines** (Version 4)

Instructions:\*

- 1. Record answers in "item response" column. If missing, mark with an X
- 2. Perform reversals as indicated, and sum individual items to obtain a score.
- 3. Multiply the sum of the item scores by the number of items in the subscale, then divide by the number of items answered. This produces the subscale score.
- 4. Add subscale scores to derive total FACT-G score.
- 5. The higher the score, the better the QOL.

| <b>Subscale</b> | Item Code | Reverse | e item? | Item response | <b>Item Score</b> |
|---|---|---|---|---|---|
| PHYSICAL | GP1 | 4 | - | | = |
| WELL-BEING | GP2 | 4 | - | | = |
| (PWB) | GP3 | 4 | - | | = |
| | GP4 | 4 | - | | = |
| Score range: 0-28 | GP5 | 4 | - | | = |
| G | GP6 | 4 | - | | = |
| | GP7 | 4 | - | | = |

Sum individual item scores: \_\_\_\_\_

Multiply by 7: \_\_\_\_\_

Divide by number of items answered: =PWB subscale

| S | c | 0 | r | e |
|---|---|---|---|---|

| <b>Subscale</b> | <b>Item Code</b> | Reverse | e item? | Item response | <b>Item Score</b> |
|---|---|---|---|---|---|
| SOCIAL/FAMILY | GS1 | 0 | + | | = |
| WELL-BEING | GS2 | 0 | + | | = |
| (SWB) | GS3 | 0 | + | | = |
| | GS4 | 0 | + | | = |
| Score range: 0-28 | GS5 | 0 | + | | = |
| score range. 0 20 | GS6 | 0 | + | | = |
| | GS7 | 0 | + | | = |

Sum individual item scores: \_\_\_\_\_

Multiply by 7: \_\_\_\_\_\_\_

Divide by number of items answered: \_\_\_\_\_\_=SWB subscale

| • | n | ^ | | ^ |
|---|---|---|---|---|
| Э | u | u | ı | C |

| <b>Subscale</b> | <b>Item Code</b> | Item Code Reverse item? | | Item response | <b>Item Score</b> |
|---|---|---|---|---|---|
| <b>EMOTIONAL</b> | GE1 | 4 | - | | = |
| WELL-BEING | GE2 | 0 | + | | = |
| (EWB) | GE3 | 4 | - | | = |
| | GE4 | 4 | - | | = |
| Score range: 0-24 | GE5 | 4 | - | | = |
| | GE6 | 4 | _ | | = |

| | | Sum individual item scores: | | | | |
|---|---|---|---|---|---|---|
| | | | | | Multiply by 6: | |
| Divide | | | by number of items an | | | |
| score | | | | .,, | | |
| Subscale | <b>Item Code</b> | Rever | se item? | Item response | Item Score | |
| FUNCTIONAL | GF1 | 0 | + | <del></del> | = | |
| WELL-BEING | GF2 | 0 | + | | = | |
| (FWB) | GF3 | 0 | + | | = | |
| , | GF4 | 0 | + | | = | |
| G 0.20 | GF5 | 0 | + | | = | |
| Score range: 0-28 | GF6 | 0 | + | | = | |
| | GF7 | 0 | + | | = | |
| | Sum individual item scores: | | | | | |
| | | Multiply by 7: | | | | |
| | | | Divide | by number of items an | | =FWB subscale |
| score | | | | , , | | |
| <b>Subscale</b> | Item Code I | Reverse | item? | Item response | Item Score | <u>e</u> |
| THROMBO- | An5 | 0 | + | | = | |
| CYTOPENIA | An7 | 0 | + | | = | |
| SUBSCALE | Th1 | 4 | - | | = | |
| (ThS) | Th2 | 4 | - | | = | |
| | Th3 | 4 | - | | = | |
| | Th4 | 4 | - | | = | |
| Score range: 0-72 | Th5 | 4 | = | | = | |
| | Th6 | 4 | = | | = | |
| | Th7 | 4 | = | | = | |
| | Th8 | 4 | - | | = | |
| | Th9 | 4 | - | | = | |
| | HI7 | 4 | - | | = | |
| | Th10 | 4 | - | | = | |
| | Th11 | 4 | - | | = | |
| | Th12 | 4 | - | <del></del> | = | |
| | Th13 | 4 | - | <del></del> | = | |
| | Th14 | 4 | - | | = | |
| | Th15 | 4 | - | | = | |
| | | Sum individual item scores: | | | | |
| | | | y by 18: | | | |
| | | | Divide b | y number of items answ | vered: | = <u>Th Subscale</u> |
| score | | | | | | |
| To derive a FACT- | I'h Trial Outcome | Index ( | TOI): | | | |
| Score range: 0-128 | | | | | | |
| | | _ | | | =: | = <u>FACT-Th TOI</u> |
| | | (F | PWB score | ) (FWB score) (ThS s | score) | |

| To Derive a FACT-G | total score: | | | | | |
|---|---|---|---|---|---|---|
| Score range: 0-108 | | | | | | |
| | | + | + | + | = | = <u>FACT-G Total</u> |
| | score | | | | | |
| | (PWB | score) (SWE | score) (EW | B score) (FWI | B score) | |
| | ` | | | | , | |
| To Derive a FACT-TI | n total score: | | | | | |
| Score range: 0-180 | | | | | | |
| | + | + | + | + | = | = <b>FACT-Th</b> |
| Total score | | | | | | |
| (PWI | B score) (SWB | score) (EWB | score) (FWB | score) (ThS | score) | |

<sup>\*</sup>For guidelines on handling missing data and scoring options, please refer to the Administration and Scoring Guidelines in the manual or on-line at www facit.org.